CLINICAL TRIAL: NCT06142825
Title: Developing, Implementing and Evaluating Effective Community-facility Interactions to Improve Blood Availability and Transfusion in Three Distinct County Settings in Kenya (CoBAnK): A Type III Hybrid Effectiveness-implementation Trial.
Brief Title: Developing, Implementing and Evaluating Effective Community-facility Interactions to Improve Blood Availability and Transfusion in Three Distinct County Settings in Kenya
Acronym: CoBAnK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Strathmore University (Other); University of Pittsburgh (Other); Center for Public Health and Development, Kenya (CPHD) (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B09; 5UH3HL151595-04 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Blood Transfusion

STUDY DESIGN:
Intervention Model Description: Type III hybrid effectiveness-implementation trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CFTC (Experimental): Community-Facility Transfusion Committees (CFTCs) will be established at the facilities randomized to this arm.
  Interventions: Other: Community-Facility Transfusion Committee (CFTC)
- Control (No Intervention)

INTERVENTIONS:
Other: Community-Facility Transfusion Committee (CFTC) — Community-Facility Transfusion Committees (CFTCs) are intended to incorporate diverse representation involving hospital, community, and county leadership, to improve blood availability and transfusion at the point-of-care.
  Arms: CFTC

SUMMARY:
The strategy of the CoBAnK study is to establish and enable the function of Community-Facility Transfusion Committees (CFTCs) incorporating diverse representation involving hospital, community, and county leadership, to improve blood availability and transfusion at the point-of-care.

DETAILED DESCRIPTION:
The strategy of the CoBAnK study is to establish and enable the function of Community-Facility Transfusion Committees (CFTCs) incorporating diverse representation involving hospital, community, and county leadership, to improve blood availability and transfusion at the point-of-care. The CFTC strategy will be evaluated across nine transfusing facilities across three counties in Kenya (two intervention and one control site in each county). While the intervention will be tested in "beta" facilities (i.e., facilities without a co-located blood bank) in each county, blood availability will also be measured in "alpha" facilities (i.e., facilities with co-located blood banks) in the three counties, which supply blood to the beta facilities.

ELIGIBILITY:
Eligibility criteria for study sites (beta hospitals):

* Transfusing hospital at level 3 or higher
* Has conducted at least 20 blood transfusions in the preceding year
* Does not have a KTTA-approved blood bank (regional or satellite) in the facility premises
* Receives blood from a blood bank at an Alpha Facility in the same county

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Met blood need | The time required for the hospital laboratory to process a request for blood for transfusion, up to two weeks.
  The proportion of transfusion requests resulting in dispatch of blood products from the laboratory

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
The BLOODSAFE project is committed to quickly sharing results and data. Papers will be submitted summarizing the primary results of the BLOODSAFE studies once the analysis is complete. These results will be published in major scientific journals and presented at scientific meetings.